CLINICAL TRIAL: NCT06689189
Title: Metabolite Fluorescence Analysis in Critically Ill Patients' Blood and the Development of a Blood Fluorescence Analytical Platform
Brief Title: Detection of Sepsis Occurrence by Using Blood Fluorescence
Status: Recruiting | Type: Observational
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Collaborators: University of Macau (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023SL338-01
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Sepsis; Organ Damage
Keywords: Sepsis; Organ damage; Blood metabolite fluorescence; Machine learning; Deep learning; Fluorescence spectrum analytical platform
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy control group: Individuals who are physically healthy with no underlying diseases and have not been hospitalized within the past two years. Recruitment for healthy volunteers will be conducted through notices and online media.
  Interventions: Other: Blood fluorescence metabolite analysis
- Infected Non-Sepsis Patient Group: Patients with infections and a SOFA score of 1 will be screened and confirmed by a physician to meet the inclusion criteria. After obtaining informed consent, a nurse will collect a 4 cc blood sample within 24 hours of qualification. Within 7 days of ICU admission, physicians will assess whether patients with non-sepsis infections progress to sepsis. If so, these patients will be categorized into the sepsis patient group. One week post-discharge and on the 28th day post-diagnosis, a nurse will follow up to inquire about their health status.
  Interventions: Other: Blood fluorescence metabolite analysis
- Vasopressorin treated sepsis group: Patients with confirmed infections, having qSOFA ≥ 2 and SOFA ≥ 2, accepted with vasopressor therapy, will be screened and confirmed by a physician to meet the inclusion criteria. After physician confirmation that the inclusion criteria are met, patients will be informed and asked to sign an informed consent form. Blood samples (4 cc) will be collected within 24 hours before and after hospitalization entry and within 24h after transferred out of the ICU.
  Interventions: Other: Blood fluorescence metabolite analysis
- No vasopressor theapy sepsis group: Group/Cohort Description: Patients with confirmed infections, having qSOFA ≥ 2 and SOFA ≥ 2, without vasopressor therapy, will be screened and confirmed by a physician to meet the inclusion criteria. After physician confirmation that the inclusion criteria are met, patients will be informed and asked to sign an informed consent form. Blood samples (4 cc) will be collected within 24 hours before and after hospitalization entry.
  Interventions: Other: Blood fluorescence metabolite analysis

INTERVENTIONS:
Other: Blood fluorescence metabolite analysis — This is an observational study and does not involve intervention. In both the early and late stages of sepsis, a significant increase in inflammatory free radicals changes the optical properties of the patient's blood, distinguishing it from that of healthy individuals. To explore this phenomenon, 4 cc of fasting blood is drawn from patients who pass our screening criteria. This sample is then centrifuged in accordance with our detailed standard operating procedures to ready it for analysis. Subsequently, the fluorescence intensity of the blood is measured quantitatively using a precisely calibrated blood fluorometer, which is specifically designed to detect subtle variations indicative of both early and late sepsis. This entire process is executed under stringent quality control protocols to ensure the reliability and accuracy of the results, which are pivotal for the timely diagnosis and intervention in septic patients.

SUMMARY:
This study adopted a case-control study method to explore a reagent-free, highly sensitive, and frequently screened blood fluorescence metabolite analyzer for sepsis, which can detect the emergence of inflammatory free radicals before organ damage and shorten the diagnosis time of sepsis.

DETAILED DESCRIPTION:
Currently, clinical practice lacks an effective screening method for early detection and prediction of sepsis. This gap hinders timely differential diagnosis, leading to severe shock and increased mortality rates. Although the qSOFA score is highly specific, it is not devoid of false negatives. Typically, by the time sepsis is confirmed using the qSOFA (≥ 2) and SOFA (≥ 2) scores as gold standards, the patient may already be suffering from organ damage, thus escalating the risk of death. Early-stage septic patients exhibit a surge in inflammatory free radicals, altering the optical characteristics of their blood compared to that of healthy individuals. Based on this, we hypothesize that a blood fluorometer could detect these early changes in septic patients, enabling rapid and accurate diagnosis to mitigate mortality rates. This study will conduct a case-control investigation, collecting blood from both admitted and discharged patients, with the aim of developing a reagent-free, highly sensitive blood fluorescence metabolite analyzer. This device will be capable of frequent sepsis screenings, detecting inflammatory free radicals before organ damage occurs, thereby reducing the time to sepsis diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy control group: Individuals who are physically healthy with no underlying diseases and have not been hospitalized within the past two years. Recruitment for healthy volunteers will be conducted through notices and online media.
2. Sepsis Experimental Group: Patients with confirmed infections, having qSOFA ≥ 2 and SOFA ≥ 2, will be screened and confirmed by a physician to meet the inclusion criteria.
3. Non-septic Severe Control Group: Patients with suspected or confirmed infections, having a SOFA score of 1, will be screened and confirmed by a physician to meet the inclusion criteria.

Exclusion Criteria: minors, pregnant, individuals with mental illnesses, and other vulnerable groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy control group: Individuals who are physically healthy with no underlying diseases and have not been hospitalized within the past two years. Recruitment for healthy volunteers will be conducted through notices and online media.
  2. Sepsis Experimental Groups: Inpatients with confirmed infections, having qSOFA ≥ 2 and SOFA ≥ 2, will be screened and confirmed by a physician to meet the inclusion criteria. The experimental group in this study was divided into two subgroups. One was the group of sepsis patients who used vasopressors, and the other was the group of sepsis patients who did not use vasopressors.
  3. Non-septic Severe Control Group: Inpatients with suspected or confirmed infections, having a SOFA score of 1, will be screened and confirmed by a physician to meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
specificity and sensitivity of blood fluorescence intensity in diagnosing sepsis. | 1 year
  The primary outcome variable for this clinical trial is the specificity and sensitivity of blood fluorescence intensity in diagnosing sepsis.

SECONDARY OUTCOMES:
the correlation coefficients between the fluorescence intensity and other variables | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Institute of Innovation for Combined Medicine and Engineering (NIIME), Ningbo Medical Center Lihuili Hospital, Ningbo University, Ningbo, Zhejiang, China

REFERENCES:
- [Result] Guo F, Zhu X, Wu Z, Zhu L, Wu J, Zhang F. Clinical applications of machine learning in the survival prediction and classification of sepsis: coagulation and heparin usage matter. J Transl Med. 2022 Jun 11;20(1):265. doi: 10.1186/s12967-022-03469-6. PMID 35690822
- [Result] Li Y, He Y, Miao K, Zheng Y, Deng C, Liu TM. Imaging of macrophage mitochondria dynamics in vivo reveals cellular activation phenotype for diagnosis. Theranostics. 2020 Feb 3;10(7):2897-2917. doi: 10.7150/thno.40495. eCollection 2020. PMID 32194843
- [Result] Shen YF, Tsai MR, Chen SC, Leung YS, Hsieh CT, Chen YS, Huang FL, Obena RP, Zulueta MM, Huang HY, Lee WJ, Tang KC, Kung CT, Chen MH, Shieh DB, Chen YJ, Liu TM, Chou PT, Sun CK. Imaging Endogenous Bilirubins with Two-Photon Fluorescence of Bilirubin Dimers. Anal Chem. 2015 Aug 4;87(15):7575-82. doi: 10.1021/acs.analchem.5b01903. Epub 2015 Jul 16. PMID 26146882
- [Result] Wu X, Guo LZ, Liu YH, Liu YC, Yang PL, Leung YS, Tai HC, Wang TD, Lin JC, Lai CL, Chuang YH, Lin CH, Chou PT, Lai IR, Liu TM. Plasma riboflavin fluorescence as a diagnostic marker of mesenteric ischemia-reperfusion injury in rats. Thromb Res. 2023 Mar;223:146-154. doi: 10.1016/j.thromres.2023.01.032. Epub 2023 Feb 3. PMID 36753876